CLINICAL TRIAL: NCT05076240
Title: Impact of the FilmArray® Test on the Management of Ventilator Associated Pneumonia in COVID-19 ARDS
Brief Title: FilmArray® and Management of Ventilator Associated Pneumonia in COVID-19 ARDS
Acronym: COVIDARRAY
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2021/LD-01
Record Dates: First submitted 2021-10-08; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: SARS-CoV2 Infection; Ventilator Associated Pneumonia; Ards; COVID-19
Keywords: FilmARRAY; ARDS; COVID 19; ventilator associated pneumonia; DIAGNOSTIC
MeSH Terms: conditions — COVID-19; Pneumonia, Ventilator-Associated; Acute Lung Injury; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with ventilator associated pneumonia in COVID-19 ARDS: Patient hospitalized in intensive care unit for acute respiratory distress related to a Sars-Cov2 infection having contracted ventilator associated pneumonia. The diagnosis was made by culture but also with a FilmArray® multiplex PCR analysis.
  Interventions: Procedure: FilmArray® analysis

INTERVENTIONS:
Procedure: FilmArray® analysis — FilmArray® multiplex PCR analysis to diagnose ventilator associated pneumonia in COVID-19 ARDS

SUMMARY:
Ventilator Associated Pneumonia (VAPs) are a very common side effect in intensive care units. They are the leading causes of nosocomial infections and excess mortality in intensive care units: associated with a controversial death rate of around 13%.

VAPs complicate about 40-50% of COVID-19 acute respiratory distress syndrome (ARDS) and the mortality would be twice higher.

Thus, in this context of the COVID-19 pandemic, this represents a considerable rate of patients.

Unfortunately, the risk factors for VAPs are poorly understood and the bacterial ecology varies around the world. Also, facing a high prevalence of multi-resistant bacteria in this population, the choice of probabilistic antibiotic therapy is complex and represents a considerable impact for care.

New microbiological rapid diagnostic techniques have appeared in recent years, among them the FilmArray® seems to present interesting diagnostic performances with the ability to detects resistance to antibiotics.

This technique has been studied in acute community pneumonia but has not been validated in VAP and even less during the COVID-19 period.

Investigators decide to conduct this study to investigate if the early identification of the pathogens and their mechanism of resistance using FilmArray® would improve the relevance of the antibiotic treatment.

The aim of this project is to evaluate the contribution of a rapid diagnostic technique to the management of Ventilator Associated Pneumonia during COVID-19 acute respiratory distress syndrome before an interventional study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 yers
* COVID-19 acute respiratory distress syndrome hospitalization
* affected Ventilator Associated Pneumonia
* having multiplex PCR analysis FilmArray®

Exclusion Criteria : Patient opposition to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of 18 years old and more, hospitalized in intensive care between 27th March 2020 and April 2021 for COVID-19 acute respiratory distress syndrome, declaring a Ventilator Associated Pneumonia diagnosed by culture and having multiplex PCR analysis FilmArray®.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2021-03-27 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Impact of FilmArray® on the adaptation of antibiotic therapy | Day 7
  Proportion of patients for whom the FilmArray® technique induces an adaptation of antibiotic therapy

SECONDARY OUTCOMES:
Diagnostic Performance | Day 7
  Diagnostic performance of FilmArray® in ventilator-associated pneumonia during severe acute respiratory syndrome related to COVID 19 (evaluated by FilmArray®-culture diagnostic concordance
Bacterial ecology | Day 7
  Description of the bacterial species and proportions in ventilator-associated pneumonia during severe acute respiratory syndrome related to COVID-19
Fungal ecology | Day 7
  Description of the fungal species and proportions in ventilator-associated pneumonia during severe acute respiratory syndrome related to COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Claire ROGER, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

IPD SHARING:
Plan to Share IPD: No